CLINICAL TRIAL: NCT06950177
Title: A Phase I, Dose-escalation Study to Assess the Safety, Reactogenicity, and Immunogenicity of Two Doses of an Adjuvanted Novel Pancoronavirus Vaccine (Cov- RBD-scNP-001) in 18 Through 55-year-old Healthy Participants
Brief Title: Pancoronavirus Vaccine Study in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Pro00117785
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-04

CONDITIONS: COVID-19 Respiratory Infection; SARS CoV 2 Infection; COVID-19 Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): Participants in the Low Dose Group will receive CoV-RBD-scNP-001 50 mcg + 3M-052-AF 5 mcg intravenously at Days 1 and 29.
  Interventions: Biological: CoV-RBD-scNP-001 and 3M-052-AF
- Medium Dose (Experimental): Participants in the Medium Dose Group will receive CoV-RBD-scNP-001 100 mcg + 3M-052-AF 5 mcg intravenously at Days 1 and 29.
  Interventions: Biological: CoV-RBD-scNP-001 and 3M-052-AF
- High Dose (Experimental): Participants in the High Dose Group will receive CoV-RBD-scNP-001 150 mcg + 3M-052-AF 5 mcg intravenously at Days 1 and 29.
  Interventions: Biological: CoV-RBD-scNP-001 and 3M-052-AF

INTERVENTIONS:
Biological: CoV-RBD-scNP-001 and 3M-052-AF — All subjects will receive the investigational vaccine CoV-RBD-scNP-001 adjuvanted with 3M-052-AF.

SUMMARY:
Coronaviruses (CoVs) have caused the severe acute respiratory syndrome (SARS) outbreak, the Middle East Respiratory Syndrome (MERS) outbreak, and now the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic. Although there are several approved or authorized vaccines for SARS-CoV-2, there are currently no vaccines approved to prevent diseases caused by multiple different coronaviruses. Two countermeasures with promise for controlling coronavirus outbreaks are recombinant neutralizing antibodies and vaccines directed against the virus. Between these two countermeasures, the ultimate solution to control the current COVID-19 pandemic and future CoV outbreaks is a pancoronavirus vaccine. In particular, a vaccine that can induce broader protection and can prevent severe disease caused by current SARS-CoV-2 variants of concern would help mitigate significant morbidity and mortality following SARS-CoV-2 infection. Additionally, an optimal pancoronavirus vaccine would prevent severe disease from other SARS-related viruses in the genus of coronaviruses-betacoronavirus-that are responsible for past outbreaks or could cause the next major outbreak in humans. Such a broadly active coronavirus vaccine would be an impactful first step towards preventing all life-threatening coronavirus human disease.

The proposed vaccine immunogen (Cov-RBD-scNP-001) is composed of an engineered receptor binding domain (RBD) of SARS-CoV-2 WA-1 covalently linked in vitro to the surface of a Helicobacter pylori ferritin protein nanoparticle (RBD-scNP). The RBD has been engineered at two sites to improve its expression. The protein nanoparticle is composed of 24 individual ferritin subunits each of which can have a SARS-CoV-2 WA-1 RBD attached to it via a nine amino acid linker. The protein nanoparticle will be delivered with 3M-052-AF adjuvant - a TLR 7/8 agonist.

DETAILED DESCRIPTION:
This is a single-site Phase I clinical trial in up to 51 males and non-pregnant, non-lactating women, 18 to 55 years old, inclusive, who are in good health and meet all eligibility criteria. The clinical trial is designed to assess the safety, reactogenicity and immunogenicity of two doses, one each, administered on Days 1 and 29 of the Cov-RBD-scNP-001 vaccine administered at three dosage levels - a 50 mcg (Low Dose Cohort) followed by a 100 mcg (Medium Dose Cohort) and lastly a 150 mcg (High Dose Cohort).

Participants will be sequentially enrolled in the Low Dose, Medium Dose, and High Dose Cohorts. Within each dose cohort will be sentinel and expanded subgroups. Four participants will be enrolled into the sentinel subgroup and 13 will be enrolled in the expanded subgroup. The estimated time to complete enrollment is 6 months. The total duration of participant participation is up to 14 months.

Follow-up study visits will occur at 3 days and at 1, 2 and 4 weeks after each vaccination, as well as 6 and 12 months after the last vaccination. Solicited adverse events will be assessed for 7 days following each vaccination. Unsolicited events will be assessed for 28 days following each vaccination. Blood and mucosal samples will be obtained for safety and immunogenicity assays at select study visits. Adverse events of special interest (AESIs), Serious adverse events (SAEs), Medically attended adverse events (MAAEs), New onset chronic medical conditions (NOCMCs), and potential immune-mediated medical conditions will be collected from the first vaccination through 12 months after the last vaccination. Clinical safety laboratory evaluations will be performed prior to, and 7 days post each vaccination and 28 days following the second vaccination.

Nasal swabs will be self-collected or collected by staff at unscheduled illness visits to evaluate breakthrough SARS-CoV-2 infection (symptomatic infection or asymptomatic infection with a positive SARS-CoV-2 test outside the study).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to the initiation of any trial procedures.
2. Able to understand and agrees to comply with all planned trial procedures and be available for all study visits.
3. Male, or non-pregnant, non-breastfeeding female, age 18-55 years, inclusive, at time first study vaccination.
4. Women of childbearing potential must agree to use or have practiced true abstinence or use at least one acceptable primary form of contraception.

   Note: These criteria are applicable to females in a relationship with a male, and who are of child-bearing potential).

   Not of childbearing potential - post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, or Essure® placement).

   True abstinence is 100% of time no sexual intercourse (male's penis enters the female's vagina). (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

   Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the participant's first vaccination, tubal ligation, intrauterine devices, birth control pills, and injectable/implantable/insertable/transdermal hormonal birth control products.

   Must have used at least one acceptable primary form of contraception for at least 30 days prior to the first vaccination and continue at least one acceptable primary form of contraception through 60 days after the last vaccination.
5. Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to each study vaccination.
6. Male participants are eligible to participate if they agree to refrain from donating sperm and to be abstinent from heterosexual intercourse with a female of childbearing potential as their preferred and usual lifestyle or must agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person during the intervention period and for at least 90 days after the last dose of study product.
7. In good general health

   As determined by medical history and physical examination, including vital signs, to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of safety of participants. Chronic medical diagnoses/ conditions should be stable for the last 30 days (i.e., no hospitalizations, ER, or urgent care for condition). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis/condition in the 30 days before study vaccination Any prescription change that is due to change of health care provider, insurance company, etc., or done for financial reasons, and in the same class of medication, will not be considered a deviation of this inclusion criterion. Participants may be on chronic or as needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to participant safety or assessment of reactogenicity and immunogenicity.
8. Reported receipt of a complete primary COVID-19 vaccine series and at least one booster with last vaccination at least 16 weeks prior to study vaccine dose 1

   A complete primary COVID-19 vaccine series is defined as two Pfizer or Moderna COVID-19 vaccines.

   Booster may be either homologous or heterologous to the primary vaccine series and must be an FDA authorized/approved vaccine though authorized/approved doses may have been received as part of a clinical trial.
9. Clinical screening laboratory evaluations are within normal reference ranges or grade 1 with no clinical significance (NCS) per investigator discretion.

   Ferritin, Iron, and Total Iron Binding Capacity (TIBC)

   (White Blood Cells [WBCs] with differential, hemoglobin [Hgb], platelets [PLTs], Alanine Transaminase [ALT], Aspartate Transaminase [AST], Creatinine [Cr], Alkaline Phosphatase [ALP], Total Bilirubin [T. Bili]). ALT, AST, ALP, and creatinine values that are below the reference range will not be exclusionary as long as these values below reference range are clinically insignificant.
10. Must agree to have samples stored for secondary research.

Exclusion Criteria:

1. Positive SARS-CoV-2 PCR at screening.
2. Abnormal vital signs (Grade 1 or higher) at screening.

   Grade 1 or higher is equivalent to:

   Systolic blood pressure (SBP) ≥ 141 mmHg or ≤ 89 mmHg

   Diastolic blood pressure (DBP) ≥ 91 mmHg

   Heart rate (HR) is ≥ 101 beats per minute or ≤ 50 beats per minute

   Oral temperature ≥ 38.0°C (100.4°F)
3. Body mass index (BMI) of < 18 kilograms/square meter (kg/m^2) or > 35 kg/m^2 (inclusive) at screening
4. History of SARS-CoV-2 infection or receipt of any COVID-19 vaccine < 16 weeks prior to study vaccination.
5. Woman who is pregnant or breastfeeding.
6. Blood or plasma donation within 4 weeks prior to study vaccination.
7. Receipt of antibody or blood-derived products (except Rho D immunoglobulin) within 90 days prior to study vaccination.
8. Any self-reported or medically documented significant medical or psychiatric disease or condition(s) that, in the opinion of the site Principal Investigator (PI) or appropriate sub-investigator, precludes study participation.

   Significant medical or psychiatric conditions include but are not limited to respiratory disease (e.g., chronic obstructive pulmonary disease [COPD]) requiring daily medications currently, history of asthma in the past 5 years, or any treatment of exacerbation of an underlying respiratory disease in the last 5 years. Significant kidney disease, liver disease, or cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease), including any history of myocarditis or pericarditis, or uncontrolled cardiac arrhythmia. Neurological or neurodevelopmental conditions (e.g., history of Bell's palsy, history of four or more migraine headaches in the past 12 months that interfered with normal daily activity or any migraine headache in the past 5 years that required emergency or inpatient medical care, epilepsy, seizures in the last 5 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, transverse myelitis, stroke or transient ischemic attack, multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis, Creutzfeldt-Jakob disease, or Alzheimer's disease). Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding treated basal cell and squamous cell carcinoma of the skin, which are allowed. Any autoimmune disease, including hypothyroidism without a defined non-autoimmune cause.
9. Has an acute illness, as determined by the site PI or appropriate sub-investigator, within 72 hours prior to study vaccination.

   An acute illness that is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate subinvestigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
10. Has known human immunodeficiency virus, hepatitis B or hepatitis C infection at screening.
11. Has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus antigen or antibody at screening.
12. Has an ongoing symptomatic condition for which there are ongoing medical investigations, but no diagnosis or treatment plan.
13. Has any confirmed or suspected immunosuppressive or immunodeficient state such as asplenia, recurrent severe infections and chronic immunosuppressant medication within the past 6 months

    Chronic meaning more than 14 continuous days
14. Has taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to the first study vaccination. Intranasal, ophthalmic, or topical (skin or eyes) corticosteroids are permitted.
15. Has any significant disorder of coagulation requiring ongoing or intermittent treatment.
16. Has participated in another investigational study involving any IP within 60 days, or 5 half-lives, whichever is longer, before the first vaccine administration.
17. Has a history of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to any previous licensed or unlicensed vaccine or to the candidate vaccine components.
18. Receipt of inactivated/subunit vaccine within 14 days prior to vaccine administration or live vaccine within 28 days prior to vaccine administration.
19. Plan to receive a COVID-19 booster vaccine within the 209 days following the first study vaccination.
20. Planned international travel in the period between vaccination through Study Day 57 visit.
21. Has a history of alcohol or drug abuse within 3 years prior to study vaccination.
22. Has any diagnosis, current or past, of schizophrenia, bipolar disease or other psychiatric diagnosis that may interfere with participant compliance or safety evaluations.
23. Has been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 5 years prior to study vaccination.
24. Has a history of receipt of an investigational ferritin-based vaccine.
25. Has any abnormality or permanent body art (e.g., tattoo) that, in the opinion of the investigator, would obstruct the ability to observe local reactions at the injection site

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with solicited local and systemic reactogenicity events from the time of each study vaccination through 7 days after each study vaccination by dosage amount | Day 7, Day 36
Number of participants with study vaccine-related and unrelated unsolicited non-serious adverse events from the time of the first study vaccination through approximately 28 days after the last study vaccination (Day 57) by dosage amount | Day 57
Number of participants with clinical safety laboratory adverse events from the time of each study vaccination through approximately 28 days after each study vaccination by dosage amount | Day 29, Day 57
Number of participants with AESIs, SAEs, MAAEs, NOCMCs, and PIMMCs at any time following the first vaccination through 12 months following the last dose received by dosage amount | Day 394
  Adverse events of special interest (AESIs); serious adverse events (SAEs); medically-attended adverse events (MAAEs); new-onset chronic medical conditions (NOCMCs); potentially immune-mediated medical conditions (PIMMCs).

SECONDARY OUTCOMES:
Geometric mean ID50 titers (IU50/mL) of neutralizing antibody levels against multiple betacoronaviruses before vaccination and 28 days (Day 57) following second vaccination | Day 57
Geometric mean fold rise (ID50) titers of neutralizing antibody levels against multiple betacoronaviruses from before vaccination to 28 days (Day 57) following second vaccination | Day 57
Binding titers (BAU/mL) of antibodies to SARS-CoV-2 Spike (WA-1 isolate) protein from plasma specimens before vaccination to 28 days (Day 57) following second vaccination | Day 57

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-07-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT06950177/ICF_000.pdf